CLINICAL TRIAL: NCT01804868
Title: Efficacy of a Web Tutorial Based on Case Vignettes for Teaching Literature Critical Assessment to Nursing Students: a Randomized Controlled Trial
Brief Title: Web Tutorial Based on Case Vignettes for Teaching Literature Critical Assessment to Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RAV005
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2013-05

CONDITIONS: New Educational Technologies
Keywords: case vignette; nurse; critical assessment; randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- case vignette tutorial (Experimental): The web tutorial composed of 4 case vignettes.
  Interventions: Other: case vignette tutorial
- passive web presentation on research regulation (Active Comparator): The presentation will be a web-based voice commented video presentation on research regulation.
  Interventions: Other: passive web presentation on research regulation

INTERVENTIONS:
Other: case vignette tutorial — The web tutorial will be composed of 4 case vignettes. A case vignette is a clinical scenario based on clinical practice. It will ask a clinical problem the student will have to answer by reading a research article on a randomized clinical trial. Then he will have to answer questions about this article which are related to the major methodological points of a randomized trial. All these steps are available on a secured website.
  Other Names: case vignette tutorial for teaching literature critical appraisal to nursing students
  Arms: case vignette tutorial
Other: passive web presentation on research regulation — The presentation will be a web-based voice commented video presentation on research regulation. It will allow to preserve a minimal blinding of participants, since the participants will not be informed of the intervention evaluated and will have the opportunity to follow the other intervention after the evaluation.
  Arms: passive web presentation on research regulation

SUMMARY:
Objective: The aim of this study is to assess the efficacy of a web tutorial based on case vignettes as a complementary tool for teaching literature critical assessment to nursing students, in terms of: 1) knowledge, 2) tutorial quality and acceptability and 3) students' point of view on research participation.

Participants: Nursing second-year students from 3 universities in Paris (Paris Descartes University, Paris Diderot University and Paris 13 Nord).

Design: A randomized controlled trial will assess the teaching efficacy of a case vignettes based tutorial compared to no tutorial. In order to preserve a minimal blinding of participants, the comparator will be a basic passive teaching presentation on internet. The students will be randomized in two parallel groups. They will be evaluated on a final case vignette, and will be invited to follow the other intervention after evaluation. The allocation of participants will be done by a computerized randomization list, the sequence will be created by an independent statistician with a ratio 1: 1: 1. Since the students follow courses in different nursing institutes for each university which may have different teaching content and organization, the randomization will be stratified by nursing institute. Allocation concealment will be provided because only the statistician will have access to the randomization list. All the participants will receive an individual mail linking them to his group dedicated website. In order to preserve a minimal blinding of participants, the comparator will be a passive presentation and the participants will not be informed of the intervention evaluated and will have the opportunity to follow the other intervention after the evaluation. In parallel, both groups will follow normally their university courses.

Intervention: A case vignette is a clinical scenario based on clinical practice. It will ask a clinical problem the student will have to answer by reading a research article on a randomized clinical trial. Then he will have to answer questions about this article which are related to the major methodological points of a randomized trial. All these steps are available on a secure website.

Outcomes: The primary endpoint will be the student's knowledge of critical assessment of randomized controlled trials. It will be measured by students' score on an evaluation case vignette with multiple choice questionnaires. The secondary endpoints will be the quality perception and acceptance of the tutorial and if the tutorial has modified their perception of research participation. Responses will be ranged by a 5-point Likert scale.

Potential interests: This study takes place in the field of nursing universitary teaching. Nursing students have entered recently the universitary education system which enhances the nursing research, an emerging field in France.

The investigators hope that this complementary teaching tool will enhance the knowledge and participation of nurses in research.

Sample size expected: 506 participants.

DETAILED DESCRIPTION:
Statistical analysis :

Qualitatives variables will be presented with the number and percentage of participants and of missing data for each outcome. Quantitative variables will be presented with the number and percentage of participants, mean, standard deviation and range. Assymetrical variables will be presented with the median and the interquartile range.

Quantitative outcomes will be compared between groups with a Fisher test in a linear mixed model. (the fixed effect will be the allocation group and the random effect will be the nursing institute so as to take into account the similarity of the students for each institute).

Qualitative outcomes will be compared using a mixed effect logistic regression model (the fixed effect will be the allocation group and the random effect will be the nursing institute so as to take into account the similarity of the students for each institute).

The data analysis will be carried out as an 'intention-to treat analysis' in all randomized participants.

For the primary outcome, missing data will be dealt with the multiple imputation method. Sensibility analysis will be used to confirm the results for the primary outcome.

Two-tailed tests will be applied at a standard level of 5%. The statistical analysis will be performed with SAS 9.3 statistical software.

ELIGIBILITY:
Inclusion Criteria:

* second-year students who have completed teaching modules on clinical research methodology.

Exclusion Criteria:

* none.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
student's knowledge of critical assessment of randomized controlled trials | 21 days
  student's score on an evaluation case vignette with multiple choice questionnaires (range 0-25)

SECONDARY OUTCOMES:
student's quality perception of the tutorial | 21 days
  measured on a 5-point Likert scale
student's acceptance of the tutorial | 21 days
  measured on a 5-point Likert scale
Impact of the tutorial on student's perception of research participation | 21 days
  Question: "After completing this training, would you participate / recommend a close member or a patient to participate to a randomized controlled trial?' Answers will be measured on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Boutron, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Philippe Ravaud, MD, Professor, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre d'Epidémiologie Clinique, hôpital Hôtel Dieu, Assistance Publique-Hôpitaux de Paris, Paris, France